CLINICAL TRIAL: NCT06684249
Title: A Randomized Controlled Trial Comparing the Efficacy of Supratrochlear and Greater Occipital Nerve Blocks to Botulinum Toxin A in the Management of Chronic Migraine
Brief Title: Efficacy of Nerve Block Versus Botox in Chronic Migraine Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Awad Bessar, Assistant Professor of Diagnostic and Interventional Radiology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MigraineNBvsBotox
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Migraine; Chronic Migraine, Headache
Keywords: Migraine; Chronic Migraine; Nerve Block; Botulinum Toxin; Botox; Headache
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Two-group parallel design comparing nerve block injections with Botox injections in chronic migraine management.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to treatment allocation to ensure unbiased evaluation of efficacy and safety outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve Block Therapy (Experimental): Participants in this group will receive supratrochlear and greater occipital nerve injections consisting of a combination of local anesthetics and corticosteroids. Injections will be administered once every 12 weeks for a total of 6 months.
  Interventions: Procedure: Nerve Block Injections
- Botulinum Toxin A (Botox) Therapy (Active Comparator): Participants in this group will receive Botulinum toxin A (Botox) injections according to the standard PREEMPT injection protocol for chronic migraine. Injections will be administered once every 12 weeks for a total of 6 months.
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Procedure: Nerve Block Injections — This intervention involves the administration of supratrochlear and greater occipital nerve block injections. The injections consist of a mixture of local anesthetics and corticosteroids, designed to reduce the frequency and severity of migraine episodes. The procedure will be repeated every 12 weeks for a total duration of 6 months to assess the long-term efficacy and safety in managing chronic migraine.
  Other Names: Supratrochlear and Greater Occipital Nerve Block
  Arms: Nerve Block Therapy
Drug: Botulinum Toxin A — Participants in this arm will receive Botulinum toxin A injections as per the PREEMPT protocol tailored for chronic migraine treatment. The treatment involves multiple injections around the head and neck regions, administered every 12 weeks over a 6-month period. This standard approach aims to reduce migraine frequency through neuromodulation of pain pathways.
  Other Names: Botox
  Arms: Botulinum Toxin A (Botox) Therapy

SUMMARY:
The goal of this clinical trial is to determine whether nerve block injections (specifically, supratrochlear and greater occipital nerve injections) are as effective as Botulinum toxin A (Botox) injections in treating chronic migraine in adults.

The main questions it aims to answer are:

* Do nerve block injections reduce the number of monthly migraine days compared to baseline?
* Are there any differences in the frequency of migraine-related symptoms between the nerve block and Botox treatment groups?
* Which treatment leads to higher patient satisfaction and improved quality of life?

Participants in this study will:

* Receive either nerve block injections or Botox injections every 12 weeks.
* Visit the clinic once every month for follow-ups and assessments.
* Maintain a headache diary to record the frequency and severity of their migraines and any adverse effects experienced.
* Researchers will compare the outcomes of the two groups to determine if one treatment is superior in terms of efficacy and patient satisfaction.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess the comparative efficacy of supratrochlear and greater occipital nerve block injections versus Botulinum toxin A (Botox) injections in the management of chronic migraine. Chronic migraine, characterized by headaches on fifteen or more days per month, significantly impacts quality of life and productivity. Effective management strategies are crucial for improving patient outcomes.

Study Design: Participants will be randomly assigned to one of two treatment arms:

* Nerve block injections group, receiving supratrochlear and greater occipital nerve injections with a combination of local anesthetics and corticosteroids.
* Botox injections group, receiving the standard Botox treatment protocol recommended for chronic migraine.

Each participant will receive their assigned treatment once every 12 weeks for a total of 6 months.

The primary endpoint will be the reduction in the number of migraine days per month from baseline to the end of the treatment period. Secondary endpoints will include changes in migraine severity, frequency of acute medication use, patient-reported outcomes on pain and migraine-related disability, and treatment safety and tolerability.

Procedures:

* Baseline evaluation will include medical history, migraine frequency and severity assessment, and previous treatment history.
* Follow-up visits will occur monthly, with additional evaluations at the end of the treatment period.
* Participants will be asked to maintain a headache diary throughout the study period to record migraine occurrence, characteristics, and any acute medication use.

Significance: This study will provide valuable data on the efficacy of nerve block injections compared to Botox, potentially offering an alternative treatment for patients who do not respond well to Botox injections. Additionally, findings may influence clinical practice guidelines and patient management strategies for chronic migraine.

Relevance: Given the burden of chronic migraine and the variable patient response to existing therapies, exploring alternative treatments is crucial. This study addresses this need by comparing two distinct therapeutic approaches, thus contributing to personalized migraine management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Diagnosis of chronic migraine, defined as having headaches on 15 or more days per month for more than three months, with at least 8 of those days meeting criteria for migraine.
* Ability to provide informed consent and comply with study requirements.
* No changes in prophylactic migraine medications in the last 3 months.

Exclusion Criteria:

* History of allergy or hypersensitivity to local anesthetics or Botulinum toxin.
* Previous nerve block or Botox treatment within the last 6 months.
* Significant comorbid psychiatric or neurological disorders that could interfere with study participation or evaluation.
* Pregnancy or breastfeeding.
* Contraindications to either treatment as per product labels.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in Monthly Migraine Days | Baseline, 3 months, 6 months post-procedure
  The primary outcome is the reduction in the number of migraine days per month. This measure assesses the effectiveness of nerve block injections versus Botox injections in decreasing the frequency of migraine days from baseline to the end of the treatment period.

SECONDARY OUTCOMES:
Change in Migraine Severity | Baseline, 3 months, 6 months post-procedure
  Assessment of changes in the severity of migraine episodes using a Visual Analog Scale (VAS), a continuous scale ranging from 0 to 100, where 0 represents "no pain" and 100 represents "worst possible pain". This measure evaluates whether the treatment reduces the pain intensity of migraines.
Frequency of Acute Medication Use | Baseline, 3 months, 6 months post-procedure
  Evaluation of the change in the frequency of acute migraine medication use, documenting any reductions as a result of the treatment.
Patient Satisfaction and Quality of Life | Baseline, 3 months, 6 months post-procedure
  Measured using the Migraine-Specific Quality of Life Questionnaire (MSQ), this outcome assesses changes in the patient's quality of life and satisfaction with treatment.
Adverse Events | Throughout the study period (6 months)
  Monitoring and recording any adverse events associated with the treatments to evaluate safety profiles of the nerve block and Botox interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Bessar, MD, PhD, Principal Investigator — Assistant Professor of Diagnostic and Interventional Radiology, Zagazig Uni.
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) with other researchers. This decision is based on considerations related to patient confidentiality, data privacy concerns, and the absence of a current infrastructure for secure data sharing. The primary results of the study will be published in peer-reviewed journals and presented at scientific conferences, ensuring that the findings are accessible to the broader research community.